CLINICAL TRIAL: NCT03624439
Title: Evaluation of the Double-Lumen Tube Vivasight-DL vs. Standard Duble-lumen Tube in Normal and Difficult Airway Scenarios: A Prospective, Randomized, Crossover, Simulation Trial
Brief Title: Duble Lumen Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lazarski University (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Associate Professor, Lazarski University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI_2018_DL1
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Intubation;Difficult; Intubation; Difficult or Failed; Difficult Airway
Keywords: double-lumen tube; ETView; medical simulation; anesthesiologist; difficult airway

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal airway (Experimental): normal airway. the language has not been inflated. the instructor assessed the difficulty of intubation based on the Cormack - Lehane scale to the first degree
  Interventions: Device: Standard double-lumen tube; Device: Double-Lumen Tube Vivasight-DL
- Difficult airway (Experimental): dofficult airway. Difficult airways were obtained by means of language inflation using a simulator control panel, so as to obtain the degree of intubation difficulty assessed by an independent anesthesiologist to the third degree according to the Cormack-Lehane scale
  Interventions: Device: Standard double-lumen tube; Device: Double-Lumen Tube Vivasight-DL

INTERVENTIONS:
Device: Standard double-lumen tube — intubation using standard double-lumen tube with Macintosh laryngoscope
Device: Double-Lumen Tube Vivasight-DL — intubation using Double-Lumen Video Tube Vivasight-DL with Macintosh laryngoscope

SUMMARY:
Intrabronal intubation is one of the basic methods of airway protection during cardiac surgery. The use of double-lumen tubes in the implementation of a standard method based on macintosh laryngoscope may cause the prolongation of the procedure especially in the case of difficult airways. The aim of the study was to match the effectiveness of endotracheal intubation using a standard Macontosh laryngskop and a normal double-lumen tube versus the ETView DL tube.

ELIGIBILITY:
Inclusion Criteria:

* anesthesiologist or a person in the course of specialization
* consent voluntary participation in the study

Exclusion Criteria:

* refusal to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
intubation time | 1 day
  from taking of the intubation device to successful intubation

SECONDARY OUTCOMES:
time to visualize the glottis | 1 day
  time defined as the time from taking laryngoscope in hand until you obtain visualize the glottis
success of the first intubation trial | 1 day
  effectiveness of the first attempt of intubation by participants using four intubation devices
overall success rate | 1 day
  effectiveness measured during a maximum of three intubation attempts, confirmed by a single lung ventilation test
the degree of visibility of the glottis | 1 day
  The POGO score describes how much glottic opening is visible. A POGO score of 100% indicates visualization of the entire glottic opening from the anterior commissure of the vocal cords to the interarytenoid notch. A POGO score of 0% corresponds with no visualization of laryngeal structures.
Cormack - Lehane grade | 1 day
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)
ease of use | 1 day
  To access subjective opinions about the difficulty of the each intubation method, participants were asked to give a rating on a visual analogue scale (VAS) with a score from 1 (extremely easy) to 100 (extremely difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, PhD, Principal Investigator — Lazarski University; Jacek Smereka, Phd, Principal Investigator — Wroclaw Medical University
Locations (1):
- Faculty of Medicine, Lazarski University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study available from the corresponding author on request.

REFERENCES:
- [Background] Bialka S, Copik M, Rybczyk K, Owczarek A, Jedrusik E, Czyzewski D, Filipowski M, Rivas E, Ruetzler K, Szarpak L, Misiolek H. Assessment of changes of regional ventilation distribution in the lung tissue depending on the driving pressure applied during high frequency jet ventilation. BMC Anesthesiol. 2018 Jul 31;18(1):101. doi: 10.1186/s12871-018-0552-2. PMID 30064377
- [Background] Szarpak L, Kurowski A, Zasko P, Karczewska K, Czyzewski L, Bogdanski L, Adamczyk P, Truszewski Z. Double-lumen tube tracheal intubation in a manikin model using the VivaSight Double Lumen: a randomized controlled comparison with the Macintosh laryngoscope. Am J Emerg Med. 2016 Jan;34(1):103-4. doi: 10.1016/j.ajem.2015.10.018. Epub 2015 Oct 23. No abstract available. PMID 26527175